CLINICAL TRIAL: NCT02705937
Title: Early Phase Study Comparing the Effectiveness of a Dairy Product, Co-developed by Besancon University Hospital and the National School of Dairy Industry (ENIL), With the Reference Treatment Aequasyal® on Dry Mouth Symptoms in Patients Suffering From Xerostomia Caused by Psychotropic Medications.
Brief Title: Early Phase Study Comparing the Effectiveness of a Dairy Product With the Reference Treatment Aequasyal® on Dry Mouth Symptoms in Patients Suffering From Xerostomia Caused by Psychotropic Medications.
Acronym: LactoXeros
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Ecole Nationale de l'Industrie Laitière (ENIL) (Unknown); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: API/2015/65
Record Dates: First submitted 2016-02-03; First posted 2016-03-11 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Xerostomia
Keywords: xerostomia, Saliva, iatrogenic oral dryness, dairy product
MeSH Terms: conditions — Xerostomia | interventions — Dairy Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dairy product (Experimental): The product will be taken for 14 days
  Interventions: Other: Dairy product
- Aequasyal mouth spray medical device (Active Comparator): The spray will be taken for 14 days
  Interventions: Device: Aequasyal mouth spray

INTERVENTIONS:
Other: Dairy product — Dairy products are given to patients with the instruction to eat as many products as necessary to provide them with some relief (within a limit of 6 per day) for 14 days
  Arms: Dairy product
Device: Aequasyal mouth spray — The mouth spray will be used by patients as needed (according to the package leaflet) for 14 days
  Arms: Aequasyal mouth spray medical device

SUMMARY:
Dry mouth symptoms mostly occur as drug side-effects. Available products such as saliva substitutes are disappointing (bad taste, poor efficiency).

The hypothesis stems from the "empirical" observations that many patients alleviate dry mouth symptoms by the consumption of dairy products. Through its composition, the dairy product in itself provides relief for the patient, due both to its physical and biochemical properties, which could explain these observed improvements, and to elements related to the phenomena of consumption of food as an alternative to medication. In the latter case, hedonism takes on a role which has not been previously assessed. Initial work undertaken with the department of applied research at the National Dairy Industry School (ENIL) led to the prototyping of a new milk product, to qualify and adapt a product with a "health benefit" in patients suffering from xerostomia.

This dairy product has specific taste, texture and lubrication properties and will be tested in a randomized controlled cross-over study for its efficiency and acceptability versus a reference product (Aequasyal ®, Oxidized Glycerol Triester) on a group of 32 patients at Dijon and at Besançon University Hospitals.

This way of combatting xerostomia at the interface of patients' diet, such as it is proposed here, could help improve their quality of life, minimize harmful effects (infection, decay) and promote adherence to treatments which are responsible for xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients seen in the psychiatry department requiring the prescription of psychotropic drugs (antidepressants anxiolytics) for over 6 weeks
* Patients complaining of xerostomia
* Patients having not taken a palliative therapy against xerostomia for at least 2 weeks
* Patients having signed a free and informed consent form
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients suffering from psychotic illness
* Patients suffering from Sjogren's syndrome
* Patients having been treated by radiation therapy for head or neck cancer
* Patients having stopped a palliative therapy against xerostomia for less than 2 weeks
* Patients under 18
* Pregnant or Breastfeeding women
* Incapacitated adults
* Patients placed under tutorship or curatorship
* Patients under judicial protection
* Patients suffering from milk allergy or lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in mouth Dryness Score | Score measured at day 0, day 14, Day 21 and day 35
  Change (in centimeters measured on a Visual Analogue Scale) determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21

SECONDARY OUTCOMES:
Difficulty in chewing | Score measured at day 0, day 14, Day 21 and day 35
  Change (in centimeters measured on a Visual Analogue Scale) determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Difficulty in swallowing | Score measured at day 0, day 14, Day 21 and day 35
  Change (in centimeters measured on a Visual Analogue Scale) determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Difficulty in speaking | Score measured at day 0, day 14, Day 21 and day 35
  Change (in centimeters measured on a Visual Analogue Scale) determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Burning sensation | Score measured at day 0, day 14, Day 21 and day 35
  Change (in centimeters measured on a Visual Analogue Scale) determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Taste perception | Score measured at day 0, day 14, Day 21 and day 35
  Change (in centimeters measured on a Visual Analogue Scale) determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Silness-Loe Index measuring dental plaque | Measured at day 0, day 14, Day 21 and day 35
  Change determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Salivary flow | Measured at day 0, day 14, Day 21 and day 35
  Change determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21
Saliva pH | Measured at day 0, day 14, Day 21 and day 35
  Change determined between day 14 and day 0 will be compared to the change assessed between day 35 and day 21

CONTACTS AND LOCATIONS:
Overall Officials: Nazim NEKROUF, MD, Principal Investigator — Besancon University Hospital
Locations (1):
- CHU de Besancon, Besançon, France